CLINICAL TRIAL: NCT06810037
Title: The Effect of Mindfulness Practice Based on the Solution-Focused Approach on Self-Esteem, Mindfulness, and Anxiety Levels of University Students
Brief Title: Solution-Focused Mindfulness: Impact on Students' Self-Esteem, Mindfulness, and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra ERDOĞAN, Assistant Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ondokuz Mayıs University
Record Dates: First submitted 2025-01-13; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: mindfulness; Self-esteem,; solution-focused therapy; anxiety; university students
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In the study, a randomized controlled experimental study design was used in order to determine the effect of the program. The third- and fourth-year university students who volunteered to participate in the study attended the eight-week Mindfulness program based on the Solution-Focused Approach.The study group of the research consisted of third- and fourth-year students who were attending the faculty of education of a university located in the Black Sea Region of Turkiye and volunteered to participate in the study. A total of 41 students (experimental group = 21, control group = 20) participated in the study. One student in the experimental group who did not regularly attend the sessions and one student from the control group who left some items blank after checking their answers were excluded from the data set. The study was completed with a total of 39 students (experimental= 20, control= 19).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Behavioral: Mindfulness Practice Based on the Solution-Focused Approach
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness Practice Based on the Solution-Focused Approach — the experimental group received 90 minutes of solution-oriented based mindfulness practices one day a week for eight weeks
  Arms: experimental group

SUMMARY:
Students have some problems related to stress and anxiety during their university years when they go through important transitions and change processes in their lives. In this sense, mindfulness program based on solution-focused approach is considered to raise the mindfulness levels of students, reinforce their self-esteem, and lower their anxiety levels. Therefore, this study comprehensively examined the effects of mindfulness program based on solution-focused approach on the self-esteem, mindfulness levels, and anxiety of university students. A significant difference was found between the scores of the students before and after the program on their trait anxiety levels, mindfulness, and self-esteem levels. In this case, it could be asserted that the mindfulness program based on the solution-focused approach had positive effects on their self-esteem, mindfulness, and anxiety levels of the students.

ELIGIBILITY:
Inclusion Criteria:

* To be a third and fourth year student of Samsun Ondokuz Mayıs University Faculty of Education,
* Not working in a private or state institution,
* Not having a disease that prevents sitting or walking in order to be able to perform the applications,
* Having anxiety about the future (it will be questioned whether it is present in the preliminary interview)

Exclusion Criteria:

* Have a diagnosed serious physical illness or chronic disease,
* Having a diagnosed psychiatric illness,
* Having experienced the loss of a family member or loved one within the last six months,
* History of substance abuse, suicide attempt or self-harm,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Rosenberg Self-Esteem Scale (RSES) | first week and the end of the eighth week
  Morris Rosenberg (1965) developed the scale to assess self-esteem in adolescents. Çuhadaroğlu (1986) conducted the reliability and validity study of the scale in Turkiye. The scale has a total of 63 items. For the purpose of the study, the first 10 items of the scale were used to assess self-esteem. The questions are rated by the Guttman evaluation method. A score of 0-1 indicates a high level of self-esteem, 2-4 indicates a medium level of self-esteem and 5-6 indicates a low level of self-esteem

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory-STAI | first week and the end of the eighth week
  Spielberger et al., (1970) developed the State and Trait Anxiety Inventory, consisting of two subscales, each with 20 items. Öner and Le Compte (1985) adapted the State-Trait Anxiety Inventory into Turkish and conducted its validity and reliability. The State Anxiety subscale (STAI-S) determines how the individual feels at a specific moment and under certain conditions, and the Trait Anxiety subscale (STAI-T) determines how the individual usually feels. The total score for both subscales ranges between 20-80 points; high scores indicate a high level of anxiety. During the score calculation of the State Anxiety Inventory, items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 are reversed expressions. During the score calculation of the Trait Anxiety Inventory, items 21, 26, 27, 30, 33, 36, and 39 are reversed expressions
Mindful Attention Awareness Scale (MAAS) | first week and the end of the eighth week
  Brown and Ryan (2003) developed a 15-item scale to assess the general tendency to be mindful of and attentive to momentary experiences in daily life. Özyeşil et al., (2011) conducted the validity and reliability of the scale in Turkiye. The MAAS is a 6-point Likert-type scale. The MAAS has a single-factor construct and yields a single total score. High scores of the scale indicate a high level of mindfulness

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant data may be provided by researchers upon appropriate requests, taking into account the protection of personal data.